CLINICAL TRIAL: NCT06651658
Title: Pleural Blood Patch for Lung Ablation: a Randomised Trial (Oxford Pleural Embolisation Trial - OxPET)
Brief Title: Oxford Pleural Embolisation Trial
Acronym: OxPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Yan-Lin Li, Chief Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18274
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Lung Metastases
Keywords: lung cancer; lung metastases; lung ablation; pleural embolisation; Pleural blood patch
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung ablation only (No Intervention): Patients proceed to standard of care treatment with lung ablation as deemed clinically appropriate
- Lung ablation with pleural embolisation (Experimental): In addition of standard of care lung ablation, patients undergo pleural blood patch embolisation during withdrawal of the ablation probe
  Interventions: Procedure: Pleural embolisation

INTERVENTIONS:
Procedure: Pleural embolisation — Administration of pleural blood patch with tandem needle technique
  Arms: Lung ablation with pleural embolisation

SUMMARY:
Thermal ablation is an established treatment for lung cancer. It involves insertion of a applicator under image guidance into a lung tumour and destroying it with radiofrequency, microwave or cryotherapy. One of the common side effects is pneumothorax, which is a leak of gas from the lungs when it punctured. Air leak necessitates placement of a drainage tube in more than half of patients undergoing the procedure. The drain can be associated with some morbidity including pain, reduced mobility, prolonged hospital stay and infection Pleural embolization refers to the injection of substances to the linings of the lung to seal air leakage. There is published evidence in using pleural embolization with autologous blood (blood drawn up from the patient's veins) to prevent pneumothorax in patients undergoing lung biopsies. This technique is also known as pleural blood patch (PBP). A study involving more than 4000 patients found that PBP reduced the rates of pneumothorax by 35% and drain placement by 55% in lung patients. A study using prophylactic gelfoam torpedo embolization for radiofrequency ablation showed significant reduction in chest drain rates.

In this study, investigators plan to evaluate the PBP using a tandem needle technique in patients undergoing lung ablation at the Oxford Thermal Ablation Service, one of the largest units in the country performing about 200 ablations per year, mostly microwave ablations. Patients will be randomized to receive lung ablation with or without the PBP.

The PBP technique is easy to learn, enjoys high technical success rates and does not expose the patient to any significant additional risk.

The primary outcome is the chest drains rates in the two trial groups:

1. patients undergoing lung ablation without PBP and
2. patients undergoing lung ablation with PBP. Other outcomes that would be measured include the volume of gas leakage on Computed Tomography (CT) imaging, safety profile, length of stay, feasibility of same day discharge, patient oriented outcomes including validated pain score, and institution oriented outcomes including medical costs.

A positive trial could significantly reduce the side effect profile of lung ablation and hasten the patient's recovery. There could be significant savings in healthcare costs as the procedure may become safe to perform as a day procedure as opposed to an overnight procedure.

DETAILED DESCRIPTION:
Background and existing literature Image guided thermal ablation is an established treatment for lung malignancy including early stage primary cancer and oligometastases. It is a minimally invasive technique associated with rapid clinical recovery and its efficacy and safety are comparable to surgical resection and radiotherapy. It is also repeatable and feasible for patients contraindicated to other therapies, such as those with impaired lung function or interstitial fibrosis.

One of the most common side effects of lung ablation is pneumothorax, occurring in up to 67% of patients depending on definition. Clinically significant pneumothorax, typically defined as requiring perioperative insertion of chest drain, occurs in up to 58% of patients. In a local audit at Oxford University Hospitals last year, 31.7% of lung ablation patients required a chest drain.

Pleural or parenchymal tract embolisation using autologous blood (pleural blood patch/ PBP) is a recognized technique in pneumothorax prevention in image guided lung biopsies. In a meta-analysis including more than 4000 patients, drawing on mainly retrospective studies, this reduces the risk of pneumothorax by 35% and risks of chest drain by 55%.

A study using prophylactic gelfoam torpedo embolisation for radiofrequency ablation showed significant reduction in chest drain rates.

Rationale and necessity of the OxPET trial

A literature search demonstrates lack of any study examining the prophylactic use of PBP in lung ablation. There are important differences between lung biopsy and ablation that dedicated evaluation rather than direct extrapolation of results:

1. The ablation applicator is larger (at least 16G) than the biopsy needle (usually 20G).
2. The PBP technique in biopsies employ a coaxial technique which involves injection of blood along the same needle after the sample has been taken, which is not possible for ablations.
3. Ablation causes damage not just along the needle tract but a zone of destruction by thermal energy, which may render PBP ineffective.
4. Existing study using gelfoam torpedoes studied patients undergoing radiofrequency ablation and in coaxial application of embolisation agent. The majority of cases performed in OUH are with microwave technology and non coaxial application.
5. Lung ablations are performed under general anaesthesia and ventilation whereas biopsies are performed with local anaesthesia and this may cause a difference in pneumothorax formation.

The tandem needle technique is modified for PBP in the setting of ablation. This involves intraoperative CT guided insertion of a 21G needle to a position within 5mm of the parietal pleural entry of the ablation applicator. This is followed by autologous blood injection upon withdrawal of the ablation applicator. This has been evaluated clinically in selected patients at high risk of pneumothorax at OUH with promising preliminary results. We plan to publish the data as a pilot study of OxPET.

The investigation is performed at the Oxford Thermal Ablation Service, a tertiary centre performing around 200 ablations a year.

Potential clinical impact The potential clinical impact of this study is highly significant. At OUH, lung ablations are inpatient procedures requiring overnight stay, with planned discharge on the subsequent morning. Patients who require a perioperative chest drain will attempt weaning the next day, and a significant portion will fail and thus prolong discharge. A further 3.5% of patients develop drain-related complications requiring invasive management such as infection, empyema and persistent air leak, requiring further invasive management.

Significant reduction in pneumothorax rates will reduce the rate of chest drain insertion and its associated morbidities, shorten patient stay and hasten recovery. Positive trial results may shift the clinical pathway of lung ablation into a day procedure, which is increasingly the case for ablation of other organs such as the kidney.

Safety profile The PBP technique is extremely safe and no negative effects have been identified in previous meta-analysis involving more than 4000 patients. The ablation procedure would induce variable degrees of haemorrhage per se, therefore patients undergoing PBP only differs in the amount and location that the patient's blood is distributed.

There are theoretical risks of introducing infection and pneumothorax during the PBP procedure. In our protocol, a strict aseptic technique is adopted both for blood taking and ablation/ PBP procedure. A sterile surgical field is maintained and it is routine clinical practice to give a dose of prophylactic antibiotics to all ablation patients. The development of infection (pleural or pulmonary) will be monitored in our study.

With regards to pneumothorax induced by the PBP procedure, this would be immediately detected and remedied (by chest drain insertion if appropriate) as the procedure is performed under CT scanning. This complication would be recorded within the safety outcome session of the trial.

The PBP procedure is also associated with a small additional radiation exposure (0.3mSv) to intervention arm patients. The annual background radiation dose in the UK is 2.7 mSv in comparison. This has been assessed by independent medical physics and clinical radiation expert at the local institution. Opinion of the physics expert is that the additional radiation for interventional trial participants would cause a <0.01% increase in lifetime cancer risk. The opinion from the clinical radiation expert is that there is no increase in radiation exposure on a clinical level.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated for lung ablation.
* Willing and capable of giving informed consent.
* Aged 18 years or above.

Exclusion Criteria:

* Unable to proceed to lung ablation procedure.
* 3 or more lung lesions to be ablated in the same setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Perioperative chest drain insertion | (<24 hours)
  To compare the rates of clinically important pneumothorax in patients undergoing lung ablation with or without pleural blood patch embolisation
  Chest drain rates (%) are expressed in means and standard deviations.

SECONDARY OUTCOMES:
Pneumothorax volume on immediate post ablation CT imaging | Immediate post operative
  To evaluate the difference in volume of pneumothorax between intervention and control group
  Pneumothorax volume (mL) are expressed in means and standard deviations.
Technical success in interventional group | immediate post operative
  To evaluate the technical success rate of the intervention in concern
  Technical success rate (%) is only for interventional group and expressed in a descriptive percentage.
Adverse events deemed due to PBP | Through study completion, an average of 3 months
  To evaluate the safety of pleural blood patch embolisation
  Adverse event is quantified by CIRSE system (1-6), an ordinal scale variable.
Pain score | Assessed at discharge, typically day after procedure
  To evaluate the patient tolerance between intervention and control group
  Measured by visual analogue scale 1-10 ( interval scale variable, expressed in means and standard deviations)
Length of stay | Assessed at discharge, typically day after procedure
  To evaluate the patient journey between intervention and control group
  Length of stay (days): expressed in means and standard deviations.
Feasibility of same day discharge | Assessed at discharge, typically day after procedure
  To evaluate the patient journey between intervention and control group
  Feasibility of discharge at end of ablation date (yes/no): categorical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Yan-Lin Li Consultant Interventional Radiologist, EBIR FRCR FHKAM, Principal Investigator — Oxford University Hospitals NHS Foundation Trust/ University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li YL, Tan Y, Shah R, Harris V, Dmytriw A, Gleeson F, Scott S, Lyon P, Anderson EM. Tandem Needle Technique Pleural Blood Patch Embolisation for Lung Ablations. Cardiovasc Intervent Radiol. 2025 Dec 14. doi: 10.1007/s00270-025-04301-6. Online ahead of print. PMID 41392212